CLINICAL TRIAL: NCT03244332
Title: HEMOCC Study Hemostasis in Cirrhotic Children : Assessment of Risk Factors of Spontaneous Bleeding From Oesophageal Varices in Cirrhotic Children Waiting for a Graft.
Brief Title: HEMOCC Study. Hemostasis in Cirrhotic Children.
Acronym: HEMOCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013/06JUI/358
Record Dates: First submitted 2017-07-27; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Esophageal and Gastric Varices; Child, Only
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Intervention Model Description: The investigators aim to start a prospective and observational study over a 2 years period.
  First, the investigators will identify all children suffering from cirrhosis irrespective of underlying etiology and/or portal hypertension coming into the pediatric hepatogastroenterology unit at Saint-Luc University Clinics. Any patient with a congenital or acquired thrombophilia/haemorrhaegic disorder will be excluded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompensated cirrhosis (Experimental): Children suffering from decompensated cirrhosis and needing an orthotopic liver transplantation.
  Interventions: Other: Collecting Clinical Data; Other: Collecting laboratory data
- Compensated cirrhosis (Experimental): Children suffering from a compensated cirrhosis (compensated cirrhosis with kasai surgery in biliary atresia patients e.g) or from portal hypertension without cirrhosis (portal vein thrombosis e.g)
  Interventions: Other: Collecting Clinical Data; Other: Collecting laboratory data

INTERVENTIONS:
Other: Collecting Clinical Data — Clinical data as height, weight, mid upper arm circumference, jaundice, portal hypertension signs (ascites, splenomegaly, umbilical veinous circulation)
Other: Collecting laboratory data — Laboratory data as CRP, hemogram, albumin, total and conjugated bilirubin, creatinin, urea, liver enzymes, tests of hemostasis.

SUMMARY:
Prospective investigations into the role of hemostatic factors in the risk of variceal bleeding among children with chronic liver disease (thromboelastometry e.g) is still required. A better understanding of these factors would permit better risk stratification and targeted prophylaxis or therapy.

DETAILED DESCRIPTION:
The investigators aim to start a prospective and observational study over a 2 years period.

First, the investigators will identify all children suffering from cirrhosis irrespective of underlying etiology and/or portal hypertension coming into the pediatric hepatogastroenterology unit at Saint-Luc University Clinics. Any patient with a congenital or acquired thrombophilia/haemorrhagic disorder will be excluded. The investigators expect to include 20 to 30 children in the study.

The investigators will meet the parents to give them explanations about this study and its implications. Then the investigators will get the free and informed consent about the participation to this clinical study. Parents are obviously free to refuse to take part in this clinical study and to retire from it at any moment.

ELIGIBILITY:
Inclusion Criteria:

* Children suffering from decompensated cirrhosis and needing an orthotopic liver transplantation
* Children suffering from a compensated cirrhosis (compensated cirrhosis with kasai surgery in biliary atresia patients e.g) or from portal hypertension without cirrhosis (portal vein thrombosis e.g)
* Each patient will have a comprehensive assessment of portal hypertension (abdominal US-Doppler and upper gastrointestinal endoscopy) and hemostasis

Exclusion Criteria:

* No underlying disease which can alter hemostasis (hemophilia, sepsis…)
* No medication which can alter hemostasis (aspirin, anti-inflammatory drugs,…)

Ages: 4 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
To evaluate risk factors of spontaneous bleeding from oesophageal varices which are independant of liver functions | over 2 year period

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Stephenne, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan at this time

REFERENCES:
- [Derived] Bonnet N, Paul J, Helleputte T, Veyckemans F, Pirotte T, Pregardien C, Eeckhoudt S, Hermans C, Detaille T, Clapuyt P, Menten R, Dumitriu D, Reding R, Scheers I, Varma S, Smets F, Sokal E, Stephenne X. Novel insights into the assessment of risk of upper gastrointestinal bleeding in decompensated cirrhotic children. Pediatr Transplant. 2019 Jun;23(4):e13390. doi: 10.1111/petr.13390. Epub 2019 Mar 19. PMID 30888111